CLINICAL TRIAL: NCT04046523
Title: Non-Invasive and Non-Contact Intracranial Pressure Waveform Recording Using Dynamic Video Ophthalmoscopy
Acronym: ICP Waveform
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Hennepin County Medical Center, Minneapolis (Other); Minnesota Office of Higher Education (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: PEDS-2019-28052
Record Dates: First submitted 2019-07-10; First posted 2019-08-06 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Intracranial Pressure Increase
Keywords: video ophthalmoscope; intraocular pressure; electrocardiogram; photoplethysmography; retinal pulsatility; spontaneous venous pulsation; blind source separation
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Intervention Model Description: In the first phase of the experiment, a total of 20 healthy controls will test the VO device to determine which camera is the most appropriate for ICP patients and to synchronize the VO, electrocardiogram (ECG), photoplethysmography (PPG), intraocular pressure (IOP) and respiratory signals.
  The second phase of the experiment will enroll a total of 70 subjects who are undergoing ICP monitoring with a surgically placed probe will be randomly assigned into one of two groups. Each group will consist of 25 adult and 10 pediatric (aged 4-17) participants. Group A will undergo two inter-leaved examinations (up to 14 days apart). Data from the first exam will be used for SVP-ICP transfer function estimation and data from the second exam will serve for intra-group verification of the estimated transfer function. Group B participants will undergo only one examination and their data will serve as an inter-group re-test verification of the estimated transfer function.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Healthy Controls (Experimental): In the first phase of the experiment, 20 healthy controls will test the VO device to determine whether the camera with a CCD or CMOS lens is the most appropriate for use in ICP patients and to synchronize the VO, ECG, PPG, IOP and respiratory signals.
  Interventions: Device: Video ophthalmoscope
- Transfer Function Estimation (Experimental): Subjects in the second phase of the experiment (70 subjects total) will be randomized to either Group A or Group B. We anticipate that 25 adult and 10 pediatric (ages 4-17) patients will participate in each group. Individuals in Group A will have two inter-leaved examinations (1-14 days apart). Data from the first examination will serve for SVP-ICP transfer function estimation and data from the second examination will serve for the intra-group verification for the estimated transfer function.
  Interventions: Device: Video ophthalmoscope
- Intra-Group Verification (Experimental): Individuals in Group B will undergo one examination. Data from Group B participants will serve as the inter-group re-test verification of the estimated transfer function.
  Interventions: Device: Video ophthalmoscope

INTERVENTIONS:
Device: Video ophthalmoscope — Use of a custom video ophthalmoscope with either a CCD or CMOS camera lens. The healthy controls group (first 20 subjects) will provide data to help determine which lens might be best for measuring ICP patients (Groups A and B) in the second phase of the study.

SUMMARY:
This study will test the use of video ophthalmoscope to provide information about intracranial pressure without the use of invasive methods, anesthesia or contact with the eye.

DETAILED DESCRIPTION:
The monitoring of intracranial pressure (ICP) is crucial in head injuries and pathologies such as brain edema, arachnoid cyst, craniosynostosis or, in very-low-birthweight infants, post-hemorrhagic hydrocephalus. Some current methods of ICP are invasive and, in the case of lumbar puncture, require anesthesia, which can distort the measurement by 5-10 mmHg. The golden clinical standard is direct measurement using a surgically-implanted intraventricular drain connected to an external pressure transducer ("ICP probe"). However, this method carries risks such as hemorrhage, malfunction, obstruction or infection . The risk in pediatric patients is up to 5% and in adults the risk of fatal hemorrhage is 4-5% in patients with subdural and intraparenchymal monitoring devices. Due to these risks and the financial burden on patients, there have been attempts to develop tools for non-invasive ICP estimation. This study will test the use of a video ophthalmoscope that will calculate the relative waveform of intracranial pressure and provide information about intracranial compliance without the use of anesthesia, invasive methods or contact with the eye.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to sit still and fix their eyes on a target in the VO objective.
* ICP participants must have an inserted ICP probe for clinical purposes.

Exclusion Criteria:

* Diagnosis of glaucoma, retinopathy or head tremor.

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
The study will look at whether retinal video-recordings can be used to help estimate intracranial pressure. | Participants in the Healthy Control and Intra-Group Verification arms will be enrolled for one day. Transfer Function Estimation Subjects will be enrolled for up to 14 days.
  This study will help determine whether there could be a less invasive method of monitoring intracranial pressure. It is thought that the use of a video-ophthalmoscope recordings could be utilized to measure intracranial pressure. The outcome measures will be provided as z-scores.

CONTACTS AND LOCATIONS:
Overall Officials: Igor Nestrasil, MD, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No